CLINICAL TRIAL: NCT04781153
Title: The Impact of Oral Bacteria on Lung Function and Inflammation
Brief Title: Bergen Oral Respiratory Intervention Study
Acronym: BORALIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Røsland (Other)
Collaborators: European Research Council (Other); Uppsala University (Other)
Responsible Party: Sponsor-Investigator, Anders Røsland, Dentist and clinical researcher, University of Bergen
Organization: University of Bergen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #94605
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Airway Obstruction; Lung Inflammation
Keywords: Periodontitis; Oral health; Lung function; Respiratory health; Periodontal treatment; Microbiome; Oral hygiene
MeSH Terms: conditions — Periodontitis; Airway Obstruction; Pneumonia | interventions — Periodontal Index

STUDY DESIGN:
Intervention Model Description: This is a single-blinded longitudinal intervention study with two study groups. The participants will act as their own control as they enter the study with the same periodontal diagnose and receive the same periodontal treatment during the study period. The study does not aim to explore the effect of the periodontal treatment itself, but how removal of oral bacteria affects lung function. After randomization the participants in the first study arm will be moved directly into an active periodontal treatment phase including a scaling and rootplaning with adjunctive chlorhexidine. The second study arm will receive the intervention 3-4 weeks after the first study group - as a "delayed intervention group". At the first appointment they will receive prophylactic periodontal treatment and oral hygiene instructions. This will enable comparison between the immediate intervention group with the delayed intervention (oral hygiene motivation), which serves as the control group.
Who Masked: Care Provider, Investigator
Masking Description: The preventive intervention - professional tooth cleaning - cannot be blinded, but the outcome measure (lung function tests) are blinded for the operator/investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate intervention (A) (Experimental): Subjects will receive the full mouth disinfection treatment protocol (scaling and rootplaning of all periodontal pockets with adjunctive use of chlorhexidine mouthwash) immediately after baseline.
  Interventions: Procedure: Periodontal treatment
- Delayed intervention (B) (Experimental): Subjects will receive a full mouth disinfection treatment protocol (scaling and rootplaning of all periodontal pockets with adjunctive use of chlorhexidine mouthwash) 3-4 weeks after baseline. The "delayed intervention" will enable the study team to explore the effect of the participants change in behavior due to participation in a research project, and furthermore how change in oral hygiene habits might affect the lung function.
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment — Periodontal treatment (scaling and rootplaning) with adjunctive chlorhexidine use

SUMMARY:
The purpose of this study is to investigate if treatment of periodontitis (gum disease) in a relatively young and healthy population can improve lung function. It is hypothesized that removing the dental biofilm reduce the source of inflammatory bacteria that can reach the lungs, and thereby reduce lung inflammation and lead to improved lung function.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will undergo a clinical screening to determine eligibility for study entry.

The study participants will be randomized into two groups. Half of the study participants will after baseline move directly into an active periodontal treatment phase including oral hygiene instructions and professional tooth cleaning by a full mouth disinfection protocol (intervention 2). New data will be collected after 6-8 weeks of healing.

The second study group will after baseline receive prophylactic periodontal treatment by oral hygiene instructions and supragingival plaque removal (intervention 1). New data will be collected after 3-4 weeks. This group will now receive the active periodontal treatment phase (intervention 2) like the first study had initially. New data will be collected after 6-8 weeks of healing.

Both groups will receive supportive periodontal treatment every 3 months in 12 months after intervention 2.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of periodontitis (stadium I or II)
* measures of periodontal infection (PI) > 50%
* inflammation (bleeding index/bleeding on probing) > 50%
* never-smoker

Exclusion Criteria:

* asthma
* symptoms of pollen allergy
* chronic lung diseases
* daily medication use which may interfere with the evaluation of the subject
* pregnancy
* use of systemic antibiotics last six months
* subgingival scaling last six months
* regularly use of oral antiseptic mouth rinse
* use of snus (moist/smokeless tobacco)
* current medical condition which may interfere with the evaluation of the subject

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) (L) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Change in Forced vital capacity in liters (L).
Forced Expiratory Volume in one second (FEV1) (L) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Change in Forced expiratory volume in one second in liters (L).
Forced Oscillation Technique (FOT) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Change in lung function measured by Forced Oscillation Technique (FOT). Outcome parameters are: Resistance at 5Hz (R5) [kPaL-1s] Resistance at 20Hz (R20) [kPaL-1s] Reactance at 5 Hz (X5) [kPaL-1s] Reactance area AX [kPaL-1] and Resonance frequency (fres) [Hz].

SECONDARY OUTCOMES:
Sampling of plaque bacteria | Change from baseline at 6 months
  Saliva and plaque collected at inclusion and from each follow-up will be analyzed with high-throughput sequencing techniques to characterize the bacteria that are present. Bacterial DNA will be isolated from the samples and the 16S rRNA bacterial gene will be amplified and sequenced by Illumina® MiSeq platforms. Shotgun sequencing will also be applied on a subsample to allow full resolution and identification of bacteria at species and subspecies taxonomic level.
Fractional exhaled nitric oxide (FeNO) | Baseline, 3 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months
  Change in FeNO at exhalation flow-rate of 50 mL/s, measured in parts per billion (ppb).

CONTACTS AND LOCATIONS:
Overall Officials: Randi Jacobsen Bertelsen, PhD, Study Chair — University of Bergen
Locations (1):
- Department of Clinical Dentistry, University of Bergen, Bergen, BERGEN, Norway

IPD SHARING:
Plan to Share IPD: No
Due to the relatively small number of participants that will be enrolled in the present study, we cannot make individual participant data openly available. However, other researcher can contact us if they are interested in discussing the possibility of getting access to the data.

REFERENCES:
- [Derived] Rosland A, Bertelsen RJ, Heinrich J, Lie SA, Malinovschi A, Bunaes DF. Effect of periodontal therapy on lung function: a twelve-month follow-up intervention study. Respir Res. 2025 May 3;26(1):172. doi: 10.1186/s12931-025-03246-1. PMID 40319277